CLINICAL TRIAL: NCT01267747
Title: Prospective Assessment of The Prevalence of Primary Aldosteronism in Hypertensive Patients Presenting With Atrial Flutter or Fibrillation
Brief Title: Prevalence of Primary Aldosteronism in Hypertensive Patients Presenting With Atrial Flutter or Fibrillation
Acronym: PAPPHY
Status: Completed | Type: Observational
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Gian Paolo Rossi, MD, FAHA, FACC, MD, FAHA, FACC, University Hospital Padova
Other Study IDs: GPR-PAPPHY
Record Dates: First submitted 2010-12-27; First posted 2010-12-28 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Atrial Fibrillation; Atrial Flutter; Aldosteronism
Keywords: Atrial fibrillation; Atrial Flutter; Primary Aldosteronism; Aldosterone Producing Adenoma
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Hyperaldosteronism; Adrenocortical Adenoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood will be withdrawn to measure levels of ions (sodium, potassium), creatinine, and TSH in the serum, and HbA1c levels, plasma aldosterone concentration (PAC), renin concentrations (DRA) or renin activity (PRA) in the plasma.
  Urine specimens to measure microalbuminuria. Buffy coat will be stored for downstream gene analysis (next study).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Atrial fibrillation or flutter patients: Patients with 'lone' paroxysmal, persistent, or permanent atrial fibrillation

SUMMARY:
Primary objective of the PAPPHY Study is to establish the prevalence of primary aldosteronism (PA) in consecutive hypertensive patients referred for 'lone' paroxysmal, persistent or permanent atrial flutter or fibrillation (AFF).

Design: cohort multicenter prospective study. State-of-the-art criteria and guidelines were followed for case detection and management of both PA and of AF in all enrolled patients (Funder J. J Clin Endocrinol Metab 2008 and 2016; Kirchhof P. Eur Heart J 2011 and 2016).

DETAILED DESCRIPTION:
A previous retrospective study documented a 12-fold increase of the risk of AFF in patients with primary aldosteronism (PA) as compared to subjects with primary (essential) hypertension (Milliez 2005). However, being retrospective this investigation could involve a selection bias and therefore is to be regarded as hypothesis-generating rather than a proof-of-concept study.

Hence, based on results of experimental studies, we hypothesize that in a proportion of hypertensive patients presenting with 'lone' PA could be the underlying cause of hypertension leading to AFF. If proven, this hypothesis would imply that an early diagnosis of PA might not only cure PA and hypertension but also prevent AFF in a non negligible number of hypertensive patients.

Primary objective is to establish the prevalence of PA in consecutive hypertensive patients referred for 'lone' paroxysmal, persistent or permanent AFF.

Study design: Prospective multicenter cohort study.

Sample size:

Based on the PAPY study experience and on available data from the literature concerning prevalence studies, we anticipated that the enrolment of at least 1000 consecutive patients will give conclusive evidence on PA prevalence in AFF patients.

Nothwithstanding a long enrolment period (from 2015 to 2018), we were unable to reach the calculated sample size and, therefore, the study was smaller than the size calculated when the PAPPHY study was conceived. In order not to introduce a time-dependent bias associated with an unduly long recruitment with associated changes in practice, it was decided to stop the study upon screening of 411 patients.

Data analysis. Data collection in a specific software, with the database securely stored and analyzed at the core laboratory of the Arterial Hypertension Unit at the University of Padova, Italy.

Experimental Procedures.

Baseline visit

* Clinic evaluation of the patient;
* Collection of demographic data and history;
* Measurement of blood pressure and heart rate;
* Scanning and storage of ECG documenting AFF;
* Echocardiography for measurement of left atrial and aortic diameters, left ventricular thickness and diameters, systolic and diastolic and transmitral Doppler flow velocity indexes;
* Clinical chemistry including serum ions, s-Creatinine, eGFR, HbA1c, microalbuminuria, TSH;
* Measurement of PRA and plasma aldosterone concentration (PAC), under baseline and after captopril challenge, if the patient is not assuming drugs interfering with the renin angiotensin system and eventually after correction of hypokalemia;
* Cardioversion if needed.

Diagnosis of PA in patients with a florid PA phenotype, i.e. a high aldosterone to renin ratio (ARR), e.g. > 100 (in [ng *dl-1 ] * [ng *ml-1 * h-1]) with no further tests, following the Endocrine Society guidelines (Funder J. J Clin Endocrinol Metab 2016) and based on compelling evidence that in these patients the specificity approaches 100%, and the false negative rate 0% (Maiolino G. J Am Heart Assoc 2017).

Exclusion of PA when ARR < 26 and plasma aldosterone concentration (PAC) < 15 ng *dl-1 at the first or a repeated test. In all PA patients presenting with an ARR value in a grey area (i.e. between 26 and 100, and a PAC > 15 ng *dl-1) at the first and a repeated test after further 1 month wash-out, a confirmatory (captopril challenge) test to rule out false positive results (Funder J. J Clin Endocrinol Metab 2016).

At the end of this work-up, computed tomography and adrenal vein sampling in patients with biochemically confirmed PA for PA subtyping.

Diagnosis of aldosterone producing adenoma (APA) confirmed by biochemical cure, e.g. normalization of plasma renin activity (PRA) and aldosterone, after adrenalectomy.

The protocol of the study was revised in 2013 and then in 2015. Herein is reported the last approved version.

ELIGIBILITY:
Inclusion Criteria:

* Unequivocal evidence (by ECG, Holter ECG or medical charts) of AFF (paroxysmal, persistent or permanent) in patients with blood pressure > 140/90 mmHg on at least 3 office measurements, or current use of anti-hypertensive drugs;
* Written informed consent.

Exclusion Criteria:

* Patient refusal to participate to the study;
* Moderate-severe valvular or congenital or myocardial heart disease;
* Current abnormal thyroid function;
* Chronic renal failure (sCreatinine > 200 μM or eGFR < 40 ml/min, calculated with MDRD formula);
* Hemochromatosis;
* Alcohol abuse;
* Acute coronary syndrome, or history of CABG, PTCA with/without stenting, acute myocardial infarction;
* Hepatitis C virus and/or B and/or HIV infection;
* Pheochromocytoma and other known secondary forms of arterial hypertension;
* Hemodynamic instability precluding withdrawal of drugs (e.g. β-blockers, ARBs, ACE-I, diuretics), interfering with PRA (or DRA) and aldosterone measurements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertensive patients presenting with atrial fibrillation or flutter
Sampling Method: Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of PA in hypertensive patients referred for 'lone' atrial fibrillation. | 2015-2018
  Prevalence of PA in hypertensive patients referred for 'lone' paroxysmal, persistent or permanent atrial fibrillation.

CONTACTS AND LOCATIONS:
Overall Officials: Gian Paolo Rossi, MD, FAHA, Study Director — Department of Medicine -DIMED, University Hospital of Padova, Italy
Locations (1):
- Department of Medicine - DIMED, University of Padova, Italy, Padua, Italy

REFERENCES:
- [Background] Beevers DG, Brown JJ, Ferriss JB, Fraser R, Lever AF, Robertson JI, Tree M. Renal abnormalities and vascular complications in primary hyperaldosteronism. Evidence on tertiary hyperaldosteronism. Q J Med. 1976 Jul;45(179):401-10. PMID 948542
- [Background] Torio-Padron N, Huotari AM, Eisenhardt SU, Borges J, Stark GB. Comparison of pre-adipocyte yield, growth and differentiation characteristics from excised versus aspirated adipose tissue. Cells Tissues Organs. 2010;191(5):365-71. doi: 10.1159/000276594. Epub 2010 Jan 14. PMID 20090305
- [Background] Carey RM. Primary aldosteronism. Horm Res. 2009 Jan;71 Suppl 1:8-12. doi: 10.1159/000178029. Epub 2009 Jan 21. PMID 19153497
- [Background] Milliez P, Girerd X, Plouin PF, Blacher J, Safar ME, Mourad JJ. Evidence for an increased rate of cardiovascular events in patients with primary aldosteronism. J Am Coll Cardiol. 2005 Apr 19;45(8):1243-8. doi: 10.1016/j.jacc.2005.01.015. PMID 15837256
- [Background] Rossi GP, Di Bello V, Ganzaroli C, Sacchetto A, Cesari M, Bertini A, Giorgi D, Scognamiglio R, Mariani M, Pessina AC. Excess aldosterone is associated with alterations of myocardial texture in primary aldosteronism. Hypertension. 2002 Jul;40(1):23-7. doi: 10.1161/01.hyp.0000023182.68420.eb. PMID 12105133
- [Background] Rossi GP, Sacchetto A, Pavan E, Palatini P, Graniero GR, Canali C, Pessina AC. Remodeling of the left ventricle in primary aldosteronism due to Conn's adenoma. Circulation. 1997 Mar 18;95(6):1471-8. doi: 10.1161/01.cir.95.6.1471. PMID 9118515
- [Background] Watson T, Karthikeyan VJ, Lip GY, Beevers DG. Atrial fibrillation in primary aldosteronism. J Renin Angiotensin Aldosterone Syst. 2009 Dec;10(4):190-4. doi: 10.1177/1470320309342734. Epub 2009 Jul 17. PMID 19617274
- [Background] European Heart Rhythm Association; European Association for Cardio-Thoracic Surgery; Camm AJ, Kirchhof P, Lip GY, Schotten U, Savelieva I, Ernst S, Van Gelder IC, Al-Attar N, Hindricks G, Prendergast B, Heidbuchel H, Alfieri O, Angelini A, Atar D, Colonna P, De Caterina R, De Sutter J, Goette A, Gorenek B, Heldal M, Hohloser SH, Kolh P, Le Heuzey JY, Ponikowski P, Rutten FH. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). Eur Heart J. 2010 Oct;31(19):2369-429. doi: 10.1093/eurheartj/ehq278. Epub 2010 Aug 29. No abstract available. PMID 20802247
- [Background] Maiolino G, Rossitto G, Bisogni V, Cesari M, Seccia TM, Plebani M, Rossi GP; PAPY Study Investigators. Quantitative Value of Aldosterone-Renin Ratio for Detection of Aldosterone-Producing Adenoma: The Aldosterone-Renin Ratio for Primary Aldosteronism (AQUARR) Study. J Am Heart Assoc. 2017 May 21;6(5):e005574. doi: 10.1161/JAHA.117.005574. PMID 28529209
- [Background] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P; ESC Scientific Document Group. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Eur Heart J. 2016 Oct 7;37(38):2893-2962. doi: 10.1093/eurheartj/ehw210. Epub 2016 Aug 27. No abstract available. PMID 27567408
- [Background] Funder JW, Carey RM, Fardella C, Gomez-Sanchez CE, Mantero F, Stowasser M, Young WF Jr, Montori VM; Endocrine Society. Case detection, diagnosis, and treatment of patients with primary aldosteronism: an endocrine society clinical practice guideline. J Clin Endocrinol Metab. 2008 Sep;93(9):3266-81. doi: 10.1210/jc.2008-0104. Epub 2008 Jun 13. PMID 18552288
- [Derived] Seccia TM, Letizia C, Muiesan ML, Lerco S, Cesari M, Bisogni V, Petramala L, Maiolino G, Volpin R, Rossi GP. Atrial fibrillation as presenting sign of primary aldosteronism: results of the Prospective Appraisal on the Prevalence of Primary Aldosteronism in Hypertensive (PAPPHY) Study. J Hypertens. 2020 Feb;38(2):332-339. doi: 10.1097/HJH.0000000000002250. PMID 31834121